CLINICAL TRIAL: NCT04167917
Title: A Phase 1 Study of NTX-301, an Oral DNMT1 Inhibitor, in Patients With MDS and AML
Brief Title: NTX-301 in MDS/AML
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pankit Vachhani, Associate Prof of Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300004830; Southern Research (Other: Southern Research)
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NTX-301 (Experimental)
  Interventions: Drug: NTX-301

INTERVENTIONS:
Drug: NTX-301 — oral hypomethylating agent

SUMMARY:
NTX-301 is a DNMT1 inhibitor. The drug is an oral drug with preclinical data that has shown preclinical anti-leukemic efficacy. This is the first clinical trial using NTX-301 in patients with myeloid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure.
2. Men or women ≥18 years with one of the following conditions that is relapsed or refractory to at least one line of therapy:

   1. Acute myeloid leukemia as long as with myeloblast percentage in the marrow is ≤ 30% or the peripheral white blood cell count is less than 20,000 cells/μL in the absence of leukoreducing therapy (e.g., hydroxyurea, leukapheresis)
   2. MDS classified as intermediate, high, or very high risk by International Prognostic Scoring System-Revised [IPSS-R] criteria
   3. CMML classified as intermediate-2 or high risk per CMML-specific prognostic scoring system (CPSS) or clinical/molecular CPSS (CPSS-mol) criteria
3. ECOG performance status of 0, 1, or 2
4. Adequate organ function at screening defined as follows [reasonably minor changes pre-first dose are acceptable if deemed so by the investigator]:

   a) Hepatic:
   * Total bilirubin ≤2 × upper limit of normal (ULN); isolated bilirubin > 2 is acceptable if participant has a diagnosis of Gilbert's syndrome
   * Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) ≤3 × ULN.

     b) Renal:
   * estimated glomerular filtration rate (by CKD-EPI method) ≥ 40 mL/min/1.73 m2 c) Cardiac:
   * Left ventricular ejection fraction greater than 45% or the institutional lower limit of normal by either ECHO or MUGA at entry.
5. Patients must have recovered to grade 1 or less from prior toxicity or adverse events (exception of myelosuppression - neutropenia, anemia, thrombocytopenia - and alopecia). Note: Participants with treatment-related toxicities that are unlikely to resolve per the investigator may be enrolled on a case-by-case basis after discussion with the medical monitor
6. Patients must have completed any chemotherapy, radiation therapy, or biologic therapy specific to their myeloid neoplasm ≥ 2 weeks or 5 half-lives (whichever is longer)
7. Able to swallow, retain, and absorb orally administered medication
8. Expected life ≥ 4 months
9. Participants with a prior history of stem cell transplant (autologous and/or allogeneic) are allowed if all of the following are met:

   * 90 days or more have elapsed from the time of transplant
   * subject has been off systemic immunosuppressive medications (including but not limited to: cyclosporine, tacrolimus, mycophenolate mofetil, or corticosteroids) for at least 30 days prior to the first dose of NTX-301. Topical steroids are permitted
   * no signs or symptoms of acute graft versus host disease, other than Grade 1 skin involvement.
   * there are no signs or symptoms of chronic graft versus host disease requiring systemic therapy
10. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG], CTFG 2014) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. A woman is considered of childbearing potential (ie, fertile) following menarche and until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.
11. Subjects and their partners with reproductive potential must agree to use 2 highly effective contraceptive measures during the study and must agree not to become pregnant or father a child for 3 months after the last dose of study treatment. Contraceptive measures that may be considered highly effective comprise combined hormonal contraception (oral, vaginal, or transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, sexual abstinence, and surgically successful vasectomy. Abstinence is acceptable only if it is consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of birth control.

Exclusion Criteria:

1. Diagnosis or presence of any of the following:

   * acute promyelocytic leukemia
   * core-binding factor AML in first relapse
   * extramedullary leukemia
   * symptomatic or untreated Central Nervous System (CNS) disease [note that lumbar puncture (LP) is not required for study enrollment unless there is clinical suspicion for CNS disease; patients with history of CNS disease are permitted to enroll if they have previously received appropriate therapy and CNS remission has been; participants on maintenance intrathecal chemotherapy may be enrolled and continue to receive therapy]
2. Patients who are receiving any other investigational agents.
3. Pregnant women and women who are breastfeeding are excluded from this study.
4. Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to:

   * severe or uncontrolled infection
   * known HIV infection requiring protease inhibitor therapy
   * known Hepatitis B; defined as presence of hepatitis B surface antigen (HBsAg)
   * known Hepatitis C; if Hepatitis C antibody is positive, then this is defined as positive Hepatitis C RNA polymerase chain reaction (PCR) (or comparable test)
   * uncontrolled diabetes and/or hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the investigator
   * Malabsorption syndrome or other conditions that would interfere with intestinal absorption.
5. History of a second malignancy, excluding non-melanoma skin cell cancer, within the last three years. Participants with second malignancies that were indolent, in situ or definitively treated may be enrolled even if less than three years have elapsed since treatment. Consult the monitor if there are any queries.
6. History of prior solid organ transplant
7. History of prior sensitivity reaction to any cytidine derivates

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety/tolerability: Incidence of treatment related adverse events (AEs) and dose-limiting toxicities (DLTs) | 3 years

SECONDARY OUTCOMES:
Efficacy: Clinical Benefit Rate (CBR) | 3 years
  Clinical Benefit Rate (CBR), as defined as the percentage of participants achieving a complete remission (CR), complete marrow remission (mCR), partial remission (PR), stable disease (SD) lasting at least 8 weeks, or hematologic improvement (HI), per International Working Group (IWG) criteria.
Efficacy: Overall response rate (ORR) | 3 years
  Overall response rate (ORR), defined as the percentage of participants achieving a CR, mCR, or PR, per IWG criteria.
Efficacy: Progression free survival (PFS) | 3 years
  Progression free survival (PFS), defined as time from first dose to disease progression, as defined by IWG criteria, or death due to any cause, whichever occurs earlier.
Efficacy: Overall survival (OS) | 3 years
  Overall survival (OS), defined as time from first dose to death due to any cause.
Pharmacodynamics (PD): Global methylation (assay) in blood and/or marrow leukemia samples | 3 years
Pharmacokinetics (PK): Area under the curve (AUC) | 3 years
Pharmacokinetics (PK): Maximum plasma concentration (Cmax) | 3 years
Pharmacokinetics (PK): Time to reach maximum concentration (Tmax) | 3 years
Pharmacokinetics (PK): Half life (t1/2) | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Medical College of Wisconsin, Milwaukee, Wisconsin